CLINICAL TRIAL: NCT05012241
Title: The Reliability of the Nine Hole Peg Test in Patients With Multiple Sclerosis
Status: Active, not recruiting | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Kateřina Rybářová, occupational therapist, Charles University, Czech Republic
Other Study IDs: 76/21 S-IV
Record Dates: First submitted 2021-08-12; First posted 2021-08-19 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Motor Activity
Keywords: occupational therapy; fine motor skills; Nine Hole Peg Test; inter-rater reliability; variability; multiple sclerosis
MeSH Terms: conditions — Motor Activity; Multiple Sclerosis | interventions — Pain Measurement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Czech patients with multiple sclerosis: Czech patients with multiple sclerosis will be asked to fill in a questionnaire. Then they will be tested by the Nine Hole Peg Test. Video of their performance will be obtained.
  Interventions: Diagnostic Test: Nine Hole Peg Test

INTERVENTIONS:
Diagnostic Test: Nine Hole Peg Test — At first, each patient will be asked to fill in the questionnaire. Then he/she will be tested by the Nine Hole Peg Test according to the new Czech version of extended manual for this test. Audio recording of verbal instructions will be used.
  Other Names: questionnaire

SUMMARY:
The main aim of the project is to establish inter-rater reliability, internal variability and variability of results got in two different ways of the Nine Hole Peg Test administered according to the new Czech extended version manual in patients with multiple sclerosis.

DETAILED DESCRIPTION:
At least 30 patients with multiple sclerosis will be tested by Nine Hole Peg Test according to new Czech manual for this test. The testing will take place in one session. Video of patients' performance will be obtained.

The inter-rater reliability, internal variability and variability of results got in two different ways will be established.

ELIGIBILITY:
Inclusion Criteria:

* outpatients with clinically definite multiple sclerosis
* Czech language as a mother tongue
* age from 20 to 65 years
* clinically stable disease (more than 30 days since the last attack of the disease)
* Expanded Disability Status Scale (EDSS) score between 1.5-8.0

Exclusion Criteria:

* inability to complete the test attempt of the Nine Hole Peg Test
* vision impairment uncorrectable with glasses
* severe hearing loss
* inability to understand instructions
* inability to complete complete testing
* failure to sign Informed consent for the patient and Consent to the collection and processing of personal data during the study at the General University Hospital in Prague

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — based on self-representation
Study Population: Czech patients with multiple sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
results from the Nine Hole Peg Test | 10 minutes
  time in seconds and hundreds of seconds

CONTACTS AND LOCATIONS:
Locations (2):
- Czechia (2):
  - Center for Demyelinating Disease (MS center), Department of Neurology, First Faculty of Medicine, Charles University and General University Hospital in Prague, Prague
  - Department of Rehabilitation Medicine, First Faculty of Medicine, Charles University and General University Hospital in Prague, Prague

IPD SHARING:
Plan to Share IPD: No